CLINICAL TRIAL: NCT02706340
Title: Expulsion of Immediate Postplacental Copper Intrauterine Devices at Six Months: A Prospective Cohort Study (PPIUD)
Brief Title: Expulsion of Immediate Postplacental Copper Intrauterine Devices at Six Months: A Prospective Cohort Study
Acronym: PPIUD
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 822078
Record Dates: First submitted 2016-01-26; First posted 2016-03-11 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Postpartum; Intrauterine Devices, Copper

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaginal delivery: Women who have had a copper IUD placed within 10 minutes of a vaginal delivery of at least 34 weeks 0 days gestation.
  Interventions: Other: No intervention - observational study only
- Cesarean delivery: Women who have had a copper IUD placed within 10 minutes of a cesarean delivery of at least 34 weeks 0 days gestation.
  Interventions: Other: No intervention - observational study only

INTERVENTIONS:
Other: No intervention - observational study only

SUMMARY:
This is an observational study enrolling women who have had a copper intrauterine device placed immediately after childbirth. The study follows participants for 6 month in order to evaluate the primary outcome of IUD expulsion within 6 months of delivery.

DETAILED DESCRIPTION:
The purpose of the study is to measure the rate of expulsion of the copper intrauterine device (ParaGard®) when placed immediately after childbirth. Many women in the United States have unintended pregnancies. Long-acting reversible birth control methods, like the copper intrauterine device (IUD), help prevent unintended pregnancy. This is because, once in place, the copper IUD provides excellent pregnancy prevention, and women using it do not have to do anything extra to make sure it works (like taking a birth control pill every day, for example). The copper IUD is safe and well liked among women who use it. Around the world, women have been getting their IUD fitted right after childbirth for the past 20 years, and this practice has been shown to be safe. This service has been offered at HUP since early 2014. When the IUD is placed after birth, there is a chance that it could fall out, as the uterus shrinks back to its pre-pregnancy size. Women who get their IUD fitted right after childbirth will be observed, and describe the rate of IUD expulsion at 6 months postpartum. Factors associated with IUD expulsion will be noted. Adult pregnant women delivering at the Hospital of the University of Pennsylvania, desiring an immediate IUD, and willing to follow up 6 months after birth, will be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman age 18 years or more
* Pregnant, 24 weeks 0 days gestation or more OR who have had a delivery at 34 weeks 0 days gestation or more
* Anticipating a delivery at the Hospital of the University of Pennsylvania
* Desiring an immediate postplacental TCu380A IUD, OR who have given birth and received an immediate postplacental TCu380A IUD
* Able and willing to give consent in English
* Willing to follow up 6 months after delivery

Exclusion Criteria:

* Allergy or contraindication to TCu380A
* Known cervical cancer or carcinoma in situ
* History of undiagnosed abnormal vaginal bleeding prior to pregnancy
* Unwilling to follow up in the six months following delivery will be excluded

Additional exclusion criteria apply after delivery:

* Preterm delivery (33 weeks 6 days gestation or less at birth)
* Clinical diagnosis of chorioamnionitis or treatment for presumed chorioamnionitis
* No longer desiring immediate postplacental TCu380A placement
* Subjects aged less than 18 years
* Men are excluded by the nature of this women's health research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult pregnant women, at least 24 weeks' gestation, anticipating a delivery and desiring an immediate postplacental TCu380A IUD, and adult women who have had a delivery and received an immediate post placental TCu380A IUD.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to measure the rate of expulsion of the copper intrauterine device (TCu380A, marketed as ParaGard®) when placed within 10 minutes of placental delivery among women delivering at the University of Pennsylvania. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No